CLINICAL TRIAL: NCT00535639
Title: A Randomised, Multiple Dose, Dose Escalation, Double-Blind, Placebo-Controlled Phase I Study Investigating the Safety of ALK Tree Tablet in Adult Subjects With Birch Pollen Induced Rhinoconjunctivitis (With/Without Asthma).
Brief Title: Tolerability of ALK Tree Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: TT-01
Record Dates: First submitted 2007-09-25; First posted 2007-09-26 (Estimated); Last update posted 2008-02-29 (Estimated); Status verified 2008-02

CONDITIONS: Allergy
Keywords: Tolerability of ALK Tree Tablet in patients with birch pollen induced allergy
MeSH Terms: conditions — Hypersensitivity

INTERVENTIONS:
Drug: Betula Verrucosa allergen extract

SUMMARY:
This trial is performed to assess the tolerability of the ALK Tree Tablet in patients with birch pollen induced allergy

ELIGIBILITY:
Inclusion Criteria:

* A clinical history of birch pollen induced rhinoconjunctivitis (with or without mild to moderate asthma ) of at least two years prior to trial entry requiring symptomatic treatment during the birch pollen season.
* Positive Skin Prick Test response to Betula verrucosa
* Positive specific IgE against Bet v1
* FEV1 ≥ 70% of predicted value

Exclusion Criteria:

* No clinical history of perennial allergic rhinitis and/or asthma caused by an allergen to which the subject is regularly exposed and sensitised
* No clinical history of significant recurrent acute sinusitis (defined as 2 episodes per year for the last two years all of which required antibiotic treatment) or chronic sinusitis
* No conjunctivitis, rhinitis or asthma at the screening or randomisation visit
* No history of anaphylaxis, including anaphylactic food allergy, bee venom anaphylaxis, exercise anaphylaxis or drug induced anaphylaxis
* No history of angioedema

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2007-10; Primary Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Krogsgaard, MD, Principal Investigator — PhaseOne Trials
Locations (1):
- PhaseOne Trials, Hvidovre, Denmark